CLINICAL TRIAL: NCT01556113
Title: The Genetic Effect on Omega 3 Fatty Acid Supplementation for the Treatment of Non Alcoholic Fatty Liver Disease in Obese Children and Adolescents
Brief Title: Genetic Effect on Omega 3 Fatty Acids for the Treatment of Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1112009408; R01HD040787 (NIH)
Record Dates: First submitted 2012-03-12; First posted 2012-03-16 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Non Alcoholic Fatty Liver Disease; Steatohepatitis; Hypertriglyceridemia; Alanine Aminotransferase, Plasma Level of, Quantitative Trait Locus 1
Keywords: fatty liver; hypertriglyceridemia; elevated liver enzymes
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Hypertriglyceridemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- omega diet carrying CC/CG genotype (Active Comparator): Subjects homozygous for the major allele of the rs73049 SNP or heterozygous (CC and CG)
  Interventions: Other: Omega diet
- omega diet carrying GG genotype (Active Comparator): Subjects homozygous for the minor allele of the rs73049 SNP (GG)
  Interventions: Other: Omega diet

INTERVENTIONS:
Other: Omega diet — Eligible subjects will receive omega rich diet for 12 weeks with weekly appointments to obtain food records, draw serum samples and provide meals.

SUMMARY:
To explore whether there is a different response to omega-3 fatty acid rich diet with respect to the hepatic fat fraction % (HFF), triglyceride, and ALT levels between the rs738409 minor allele (GG) and the common allele homozygous (CC) of PNPLA3.

Hypothesis: We expect that subjects homozygous for the minor allele of the rs73049 SNP will lower their triglyceride, hepatic fat content, and ALT levels more with dietary intervention than the common allele homozygous supplementation.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is emerging as one of the most common complications of childhood obesity. It is associated with and predicts the metabolic syndrome, independent of overall obesity. Increased ALT levels are associated with deterioration in insulin sensitivity and glucose tolerance, as well as with increasing free fatty acid (FFA) and triglyceride levels. The prevalence of metabolic syndrome and prediabetes increases with the increases in hepatic fat content in a cohort of obese adolescents.

Fatty liver, independent of visceral and intramyocellular lipid content plays a central role in the impairment of liver, muscle and adipose insulin sensitivity in obese adolescents. Thus, fatty liver disease may be the hepatic component of the metabolic syndrome.

Omega 3 fatty acids lower plasma triglyceride concentrations. The subjects entering the omega diet study will be consuming an omega rich diet that is tailored to their caloric needs. This calculation is based on the patient's weight, age, and gender with the purpose of not modifying their weight at all. Weight maintenance is a very important factor in this arm of the study. They will be on the diet for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 10 to 19 years of age
* BMI equal or greater than the 95th percentile for age and gender
* Genotype PNPLA3 CC or GG
* Liver MRI Hepatic Fat fraction ≥5.5%

Exclusion Criteria:

* Food allergy to fish or any components of the pills which include alpha tocopherol partially hydrogenated vegetable oils including soybean oils, gelatin, glycerol, corn or iron oxide
* Pregnant or breastfeeding
* Known bleeding disorder or coagulopathy or treatment with anticoagulant mechanisms or low platelet counts, abnormal PT or PTT
* Impaired glucose tolerance, Type 1 or 2 diabetes
* Birth control pills
* Alcohol consumption
* Other liver disease
* Taking any medication that alters triglyceride levels, liver function, blood pressure, glucose or lipid metabolism
* Taking over the counter supplements that affect triglycerides or lipid metabolism including fish oil supplements
* Treatment for or diagnosis of thyroid disorder or have an elevated TSH at baseline
* Use of any antipsychotic medication
* Taking chronic anti-inflammatory medications
* Less than 100 pounds (45 kg)

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
reduction in hepatic fat fraction | 12 weeks
  subjects follow study designed meal plan

SECONDARY OUTCOMES:
reduction in triglycerides | 12 weeks
  subjects follow study designed meal plan
lower ALT levels | 12 weeks
  subjects follow study designed meal plan

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Santoro, MD/PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Name MA, Savoye M, Chick JM, Galuppo BT, Feldstein AE, Pierpont B, Johnson C, Shabanova V, Ekong U, Valentino PL, Kim G, Caprio S, Santoro N. A Low omega-6 to omega-3 PUFA Ratio (n-6:n-3 PUFA) Diet to Treat Fatty Liver Disease in Obese Youth. J Nutr. 2020 Sep 1;150(9):2314-2321. doi: 10.1093/jn/nxaa183. PMID 32652034